CLINICAL TRIAL: NCT03872726
Title: Development and Validation of a Self-reported Objective Index of Work Disability in Inflammatory Bowel Disease
Acronym: IBD-OWDI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Luigi Melcarne, Principal Investigator, Corporacion Parc Tauli
Other Study IDs: Ref.: 2019/523
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease; Disabling Disease; Disability Physical
Keywords: disability; Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background theme Crohn's disease (CD) and ulcerative colitis (UC) are chronic diseases that alternate flares of active inflammation with periods of clinical remission. The working capacity of patients may be affected both by disease activity and by the aggressive treatment or surgical intervention required for the management of the disease and its complications. Work disability and impairment are especially important in patients with inflammatory bowel disease (IBD) because the disease affects young individuals who are generally employed and fully active.

Although there are several indexes in the literature that assess the degree of work disability due to IBD, all have a high degree of subjectivity, so none can be used to request disability pensions.

Experience of the research group on the subject Our group has developed a line of research on work disability associated with IBD.

Initially the investigators have studied the parameters that condition the granting of disability pensions of Spanish courts.

Subsequently, a population study of the prevalence of work disability in Spain has been carried out.

Finally, the investigators develop and validated a disability index for CD (published in its extensive and reduced form) and for UC (currently under review).

Hypothesis The IBD generates a work disability that can be measured objectively. Establishing the parameters related to disability is essential to promote equity in administrative and judicial decisions related to the granting of disability pensions to patients with IBD.

Objective Development and validation of an objective index to measure the degree of disability in IBD.

Material and methods:

Study 1:

A self-reported and objective questionnaire of disability will be developed based on the data of the population survey already carried out by our group.

Patients from a previous study (n 293) will be included. The relationship of different objective variables and disability outcomes will be analyzed with a univariate and a subsequent multivariate analysis. Alternative work disability scores will be developed.

Study 2: for the validation of the questionnaire a new online interview will be performed, patients from patients' assocations will be asked to participate. Data Collection: patients will answer a online survey administered with the SurveyMonkey © platform.

Participant will answer questions about demographics, disease activity, treatment and complications and data regarding disability. Patients will also complete the SCDWDQ (Short Crohn's Disease Work Disability Questionnaire), Work Productivity and Activity Index (WPAI), IBDQ-9, the EuroQol and IBD-DI (IBD disability index).

Statistical analysis: psychometric properties of the index will be evaluated:

1. Convergent validity: the Spearman correlation will be used to correlate the objective disability score with IBD-DI and SCDWDQ.
2. Discriminant validity: it will be measured by the t-test among patients with different degrees of disability (inactive-active, hospitalization-no hospitalization, surgery-no surgery).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 65 years old.
* Labor assets or temporary sick leave.
* Diagnosis of IBD in the 6 months prior to the survey

Exclusion Criteria:

* Inability to understand or fill out the questionnaires.
* Refusal to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A cross-sectional observational epidemiological study will be developed by administering a survey to a large population (on a national scale in Spain) of patients with IBD occupationally active.
  Patients will be asked to complete an online survey using a form written with the SurveyMonkey © platform.
  For the validation we included more than 500 patients equally divided between CU and EC.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Development and validation of a self-reported objective index of disability in inflammatory bowel disease | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Luigi Melcarne, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Calvet X, Motos J, Montserrat A, Gallardo O, Vergara M. Analysis of court criteria for awarding disability benefits to patients with Crohn's disease. Clin Gastroenterol Hepatol. 2009 Dec;7(12):1322-7. doi: 10.1016/j.cgh.2009.01.015. Epub 2009 Feb 4. PMID 19558989
- [Background] Vergara M, Montserrat A, Casellas F, Villoria A, Suarez D, Maudsley M, Gallardo O, Ricart E, Calvet X. A new validation of the Spanish Work Productivity and Activity Impairment Questionnaire-Crohn's disease version. Value Health. 2011 Sep-Oct;14(6):859-61. doi: 10.1016/j.jval.2011.02.1179. Epub 2011 May 28. PMID 21914506
- [Background] Vergara M, Montserrat A, Casellas F, Maudsley M, Gallardo O, Ricart E, Calvet X. Validation of the Spanish Work Productivity and Activity impairment questionnaire: Crohn's disease version. Eur J Gastroenterol Hepatol. 2009 Jul;21(7):809-15. doi: 10.1097/MEG.0b013e32830f4c9e. PMID 19404204
- [Background] Ramos A, Calvet X, Sicilia B, Vergara M, Figuerola A, Motos J, Sastre A, Villoria A, Gomollon F. IBD-related work disability in the community: Prevalence, severity and predictive factors. A cross-sectional study. United European Gastroenterol J. 2015 Aug;3(4):335-42. doi: 10.1177/2050640615577532. PMID 26279841
- [Background] Vergara M, Sicilia B, Prieto L, Casellas F, Ramos A, Gomollon F, Calvet X. Development and Validation of the Short Crohn's Disease Work Disability Questionnaire. Inflamm Bowel Dis. 2016 Apr;22(4):955-62. doi: 10.1097/MIB.0000000000000678. PMID 26933747
- [Background] Ramos A, Vergara M, Melcarne L, Sicilia B, Gomollon F, Calvet X. Validation of a self-reported work disability questionnaire for ulcerative colitis. Medicine (Baltimore). 2018 Sep;97(39):e12486. doi: 10.1097/MD.0000000000012486. PMID 30278537
- [Result] Calvet X, Gallardo O, Coronas R, Casellas F, Montserrat A, Torrejon A, Vergara M, Campo R, Brullet E. Remission on thiopurinic immunomodulators normalizes quality of life and psychological status in patients with Crohn's disease. Inflamm Bowel Dis. 2006 Aug;12(8):692-6. doi: 10.1097/00054725-200608000-00004. PMID 16917223